CLINICAL TRIAL: NCT00332033
Title: Development of a Non-Invasive Treatment for Uterine Leiomyoma (Fibroids)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060029; 06-CH-0029
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-02-16

CONDITIONS: Uterine Leiomyoma; Fibroids
Keywords: Fibroids; Leiomyoma; Pirfenidone; Misoprostol; Non-Surgical; Collagen; Uterus; Uterine Fibroids; Uterine Leiomyoma
MeSH Terms: conditions — Myofibroma; Leiomyoma | interventions — pirfenidone

INTERVENTIONS:
Drug: Pirfenidone

SUMMARY:
Uterine leiomyomas (fibroids) represent a major public health problem with few effective therapies. Currently, the only definitive treatment is hysterectomy and women are demanding alternative therapies to surgery. We have developed a new approach to the treatment of uterine fibroids based on collaborative laboratory research into the molecular, ultra-structural, and histopathologic changes that occur with the transformation of normal uterine myocytes into abnormal myocytes comprising uterine fibroids. We have confirmed that excessive, dysregulated collagen production (fibrosis) and abnormal collagen deposition is an underlying etiology in the pathogenesis of leiomyoma. We will test the hypothesis that an anti-tumor drug (Pirfenidone) will decrease the size of clinically relevant leiomyomas by 30%. The specific aim is to compare the effects of pirfenidone with placebo on uterine leiomyoma volume. Thirty-two (32) women will be randomized in a double-blinded treatment design. Inclusion criteria include women that have completed child-bearing, who are candidates for hysterectomy, are using effective contraceptive, and have at least one uterine leiomyoma greater than 4 cm diameter confirmed by ultrasound. Women will be excluded if they have a body mass index greater than 33 kg/m(2), other gynecological diseases, and history of cardiovascular disease or smoking. Response in each treatment group will be assessed by T-2 weighted magnetic resonance imaging (MRI) and 3-D ultrasound imaging studies during the enrollment period. To our knowledge, this will be the first study to document the response of large fibroids to a short-term trial of an anti-tumor drug. The data will be used to further define the role of fibrosis in leiomyoma and establish other clinical trials to thoroughly evaluate such therapeutic approaches for uterine leiomyomas.

DETAILED DESCRIPTION:
Uterine leiomyomas (fibroids) represent a major public health problem with few effective therapies. Currently, the only definitive treatment is hysterectomy and women are demanding alternative therapies to surgery. We have developed a new approach to the treatment of uterine fibroids based on collaborative laboratory research into the molecular, ultra-structural, and histopathologic changes that occur with the transformation of normal uterine myocytes into abnormal myocytes comprising uterine fibroids. We have confirmed that excessive, dysregulated collagen production (fibrosis) and abnormal collagen deposition is an underlying etiology in the pathogenesis of leiomyoma. We will test the hypothesis that an anti-tumor drug (Pirfenidone) will decrease the size of clinically relevant leiomyomas by 30%. The specific aim is to compare the effects of pirfenidone with placebo on uterine leiomyoma volume. Thirty-two (32) women will be randomized in a double-blinded treatment design. Inclusion criteria include women that have completed child-bearing, who are candidates for hysterectomy, are using effective contraceptive, and have at least one uterine leiomyoma greater than 4 cm diameter confirmed by ultrasound. Women will be excluded if they have a body mass index greater than 33 kg/m(2), other gynecological diseases, and history of cardiovascular disease or smoking. Response in each treatment group will be assessed by T-2 weighted magnetic resonance imaging (MRI) and 3-D ultrasound imaging studies during the enrollment period. To our knowledge, this will be the first study to document the response of large fibroids to a short-term trial of an anti-tumor drug. The data will be used to further define the role of fibrosis in leiomyoma and establish other clinical trials to thoroughly evaluate such therapeutic approaches for uterine leiomyomas.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Parous and non-parous women who have completed child-bearing (age criteria of greater than 35 years-old, and less than 50 years-old).
* Currently practicing or willing to practice contraception throughout the duration of the study.
* Women with at least one fibroid greater than 4 cm diameter on ultrasound examination.
* Women who were planning to undergo hysterectomy for treatment of symptomatic fibroids may also participate if they are willing to defer the operation until the study is completed. The patients will understand that they may choose to have surgery or any other non-study treatment at any time after enrollment and end study participation.

EXCLUSION CRITERIA:

* Inability to comply with study visits and requirements.
* BMI greater than 33kg/m(2)
* History of a serious adverse reaction to study medication.
* Inability to tolerate MRI and 3D ultrasound procedures (i.e. presence of an intra-uterine device (IUD), pacemakers, aneurismal clips or other metallic devices that are not compatible with magnetic resonance imaging).
* Medical problems including: genetic diseases that cause fibroids, history of thromboembolic (blood clot) events or need for anticoagulation (Coumadin, Heparin, etc.).
* A history of cancer within the past 5 years.
* Abnormal liver function tests (typically, will be greater than 20% elevation). Mild elevations will be at the discretion of the investigators, but undiagnosed liver conditions will represent an exclusion criterion.
* Pregnancy or lactation. Pregnancy will be evaluated by (Beta)hCG test every 30 days. Patients will be asked to use non-hormonal contraception methods while on study drug.
* Severe anemia (hct. Less than 30). Mild anemia is common in women with fibroids.
* Recent rapid growth of fibroids (i.e. doubling in size within one-six months).
* Use any of the following medications:

  1. Oral, injectable, or inhaled steroids or megesterol within the past year
  2. Estrogen or progesterone-containing compounds (including oral contraceptives, hormone replacement therapy, transdermal/injectable/vaginal/oral preparations, herbal medications with estrogenic or anti-estrogenic effects) within the past 8-12 weeks; or GnRH analogs (Danazol) or other compounds that affect menstrual cyclicity
  3. Agents like Imidazoles, due to possible interference with metabolism.
* Unevaluated gynecologic abnormalities (unexplained vaginal bleeding, cervical dysplasia, or abnormal adnexal/ovarian mass).

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32
Dates: Start 2006-05-25; Study Completion 2007-02-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Marshall LM, Spiegelman D, Barbieri RL, Goldman MB, Manson JE, Colditz GA, Willett WC, Hunter DJ. Variation in the incidence of uterine leiomyoma among premenopausal women by age and race. Obstet Gynecol. 1997 Dec;90(6):967-73. doi: 10.1016/s0029-7844(97)00534-6. PMID 9397113